CLINICAL TRIAL: NCT00740831
Title: A Phase III, Randomised, Parallel Group, Double-blind, Double-dummy, Active Comparator-controlled, Multicenter Study to Assess the Efficacy and Safety of PGL4001 vs GnRH-agonist for Pre-operative Ttt of Symptomatic Uterine Myomas
Brief Title: PGL4001 Versus GnRH-agonist in Uterine Myomas
Acronym: PEARLII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PregLem SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGL07-022
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Results first posted 2012-11-16 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Uterine Myomas
Keywords: Uterine Myomas
MeSH Terms: interventions — ulipristal acetate; Leuprolide; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (PGL4001 5 mg) (Experimental): Drug: PGL4001 5mg (oral tablets) and leuproreline matching placebo (intramuscular injection)
  Interventions: Drug: PGL4001
- B (PGL4001 10mg) (Experimental): Drug: PGL4001 10 mg (oral tablets) and leuproreline matching placebo (intramuscular injection)
  Interventions: Drug: PGL4001
- C (GnRH-agonist) (Active Comparator): PGL4001 matching placebo (oral tablets) and leuprorelin 3.75 mg (intramuscular injection)
  Interventions: Drug: leuprorelin

INTERVENTIONS:
Drug: PGL4001 — tablets
  Other Names: Ulipristal acetate
  Arms: A (PGL4001 5 mg); B (PGL4001 10mg)
Drug: leuprorelin — solution for injection
  Other Names: GnRH-agonist
  Arms: C (GnRH-agonist)

SUMMARY:
This trial will assess the efficacy and safety of PGL4001 versus GnRH agonist, over a 3-month period for the pre-operative treatment of pre-menopausal women suffering from excessive uterine bleeding due to uterine myoma.

ELIGIBILITY:
Inclusion Criteria:

* Be a pre-menopausal woman between 18 and 50 years inclusive.
* Have excessive uterine bleeding due to myoma
* Have a myomatous uterus with at least one myoma of ≥ 3 cm diameter in size
* Be eligible for one surgical procedure: e.g. hysterectomy, myomectomy or others.
* If of childbearing potential the subject must be practicing a non-hormonal method of contraception.
* Have a Body Mass Index (BMI) ≥ 18 and ≤ 40.

Exclusion Criteria:

* Has a history of or current uterine, cervical, ovarian or breast cancer.
* Has a history of or current endometrium atypical hyperplasia or adenocarcinoma.
* Has a known severe coagulation disorder.
* Has a history of or current treatment for myoma with a Selective Progesterone Receptor Modulator (SPRM) or a GnRH-agonist.
* Has a history of or known current osteoporosis.
* Has abnormal hepatic function at study entry.
* Has a positive pregnancy test at baseline or is nursing or planning a pregnancy during the course of the study.
* Has a current (within twelve months) problem with alcohol or drug abuse.
* Is currently enrolled in an investigational drug or device study or has participated in such a study within the last 30 days.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 301 (Actual)
Dates: Start 2008-08; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Elke Bestel, Study Director — PregLem SA
Locations (46):
- Austria (4):
  - Medical University Graz, Graz
  - Medical University of Innsbruck, Innsbruck
  - Landesklinikum Thermenregion Neunkirchen; Dept. For Gynecology, Neunkirchen
  - Medical University Vienna, Vienna
- Belgium (4):
  - Hopital Erasme, Department of Obstetrics and Gynecology,, Brussels
  - Clinique Universitaire St-Luc, Brussels
  - CHR de la Citadelle, Liège
  - Clinique Universitaire de Mont-Godinne, Yvoir
- France (2):
  - Cabinet de Gynécologie Chirurgicale, Bordeaux
  - CHU de Clermont-Ferrand - Polyclinique Gynécologie-Obstétrique, Clermont-Ferrand
- Germany (8):
  - Klinik für Gynäkologie und Geburtshilfe, Chemnitz
  - Universitätsklinikum Köln Klinik und poliklinik für Frauenheilkunde und Geburtshilfe, Cologne
  - Private Practice, Frankfurt
  - Medizinische Hochschule Hannover, Frauenklinik, Abt. I für Frauenheilkunde und Geburtshilfe,, Hanover
  - Universität zu Lübeck, Klinik für Gynäkologie und Geburtshilfe, Lübeck
  - Poliklinik fur Frauenheilkunde und Geburtshilfe, Münster
  - Universitätsklinikum Tübingen, Tübingen
  - Ammerland-Klinik GmbH Frauenklinik, Westerstede
- Israel (6):
  - Soroka University Medical Center, Division of Obstetrics & Gynecology, Beersheba
  - Hadassah University Hospital, Jerusalem
  - Hadassah University Hospital, Mount Scopus, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Western Galilee Hospital Nahariya, Nahariya
  - Rabin Medical Center, Helen Schneider Hospital for Women, Petah Tikva
- Italy (7):
  - Clinica Ostetrica e Ginecologica II - Università degli Studi di Bari, Bari
  - Clinica Obstetrica - Azienda Ospedaliera Universitaria di Cagliari, Cagliari
  - Azienda Ospedaliera S. Gerardo - U. O. Ostetricia e Ginecologia, Monza
  - Policlinico Universitario Federico II, Napoli
  - Universita di Padova-Dip scienze ginecologiche e della riproduzione umana, Padua
  - Clinica Ostetrica e Ginecologica - A. O. U. Policlinico Paolo Giaccone, Palermo
  - Policlinico Universitario "Agostino Gemelli", Roma
- University Medical Center Utrecht, Gynecologist Reproductive Medicine and Surgery, Division for Reproductive Medicine, Utrecht, Netherlands
- Poland (5):
  - Prywatna Klinika Polozniczo-Ginekologiczna, Bialystok
  - INVICTA Sp. Z o.o., Gdansk
  - Private Practice, Katowice
  - Samodzielny Publiczny Szpital Klinika Ginekologii Onkologicznej i Ginekologii, Lublin
  - Gabinet Lekarski Specjalistyczny "Sonus", Warsaw
- Spain (9):
  - Institut Universitari Dexeus, Barcelona
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital Clínic i Provincial, Barcelona
  - Clínica Ginecológica CEOGA, Lugo
  - Private Practice, Madrid
  - Hospital Universitario Doce de Octubre, Madrid
  - Hospital Virgen de la Arrixaca Servicio de Ginecología Carretera Madrid-Cartagena, Murcia
  - Hospital Universitaris La Fe, Valencia
  - Hospital Universitario Dr. Peset, Valencia

REFERENCES:
- [Result] Donnez J, Tomaszewski J, Vazquez F, Bouchard P, Lemieszczuk B, Baro F, Nouri K, Selvaggi L, Sodowski K, Bestel E, Terrill P, Osterloh I, Loumaye E; PEARL II Study Group. Ulipristal acetate versus leuprolide acetate for uterine fibroids. N Engl J Med. 2012 Feb 2;366(5):421-32. doi: 10.1056/NEJMoa1103180. PMID 22296076

RESULTS

PARTICIPANT FLOW:
Groups:
- A (PGL4001 5mg): Drug: PGL4001 5mg (oral tablets) and leuproreline matching placebo (intramuscular injection)
Period: Overall Study
Arm/Group | A (PGL4001 5mg) | B (PGL4001 10mg) | C (GnRH-agonist)
Started | 97 (Safety population) | 103 (Safety population) | 101 (Safety population)
Completed | 93 (Patients who completed part A (visit 6)) | 100 (Patients who completed part A (visit 6)) | 95 (Patients who completed part A (visit 6))
Not Completed | 4 | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A (PGL4001 5mg) | B (PGL4001 10mg) | C (GnRH-agonist) | Total
Number analyzed (Participants) | 97 | 103 | 101 | 301
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 97 | 103 | 101 | 301
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 40.1 (6.2) | 40.7 (6.3) | 40.3 (6.2) | 40.3 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 103 | 101 | 301
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Austria | 8 | 12 | 8 | 28
  Belgium | 12 | 16 | 13 | 41
  Germany | 4 | 0 | 3 | 7
  Spain | 21 | 28 | 18 | 67
  Israel | 4 | 6 | 2 | 12
  Italy | 6 | 7 | 7 | 20
  Poland | 42 | 34 | 50 | 126

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Reduction of Uterine Bleeding at Week 13 Visit Defined as Pictorial Blood-loss Assessment Chart (PBAC) Score < 75 at End-of-treatment Visit (Week 13 Visit)
Description: Uterine bleeding was assessed with the use of the PBAC, a validated self-reporting method to estimate menstrual blood loss.
  Patients recorded daily the number of tampons and towels used and the degree to which individual items were soiled with blood (plus small or large clots). Monthly scores range from 0 (amenorrhea) to more than 500, with higher numbers indicating more bleeding.
  A slightly stained tampon/towel scores 1, a partially stained tampon/towel scores 5, a completely saturated tampon scores 10 and a completely saturated towel scores 20. Small clots/flooding (2cm) score 1. Large clots/flooding (3cm) score 5.
  Menorrhagia is defined as a PBAC > 100 during one menstrual period which approximates to a blood loss of > 80 mL. A PBAC of 400 corresponds to a blood loss of around 300 mL or approximately 80 tampons/towels used.
  The week 13 PBAC score was calculated using the last 28 days of treatment.
Time Frame: 3 months
Population: Per protocol
Measure: Number; unit: percentage of patients
Arm/Group | A (PGL4001 5mg) | B (PGL4001 10mg) | C (GnRH-agonist)
Number analyzed (Participants) | 93 | 95 | 92
percentage of patients | 90.3 | 97.9 | 89.1
Statistical Analysis 1: Comparison: A (PGL4001 5mg) vs C (GnRH-agonist); As comparison involved two doses of PGL4001 vs GnRH-agonist, Bonferroni correction used to adjust confidence intervals; Test type: Non-Inferiority or Equivalence — Non-inferiority analysis based on the use of one-sided confidence intervals, using 2.5% level of statistical significance; Difference in proportions = 1.2, 97.5% CI 1-sided [lower limit -9.3] — Newcombe-Wilson method for CI. Percentage in A minus percentage in C needed to be greater than non-inferiority margin of -20%
Statistical Analysis 2: Comparison: B (PGL4001 10mg) vs C (GnRH-agonist); As comparison involved two doses of PGL4001 vs GnRH-agonist, Bonferroni correction used to adjust confidence intervals; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in proportions = 8.8, 97.5% CI 1-sided [lower limit 0.4] — Newcombe-Wilson method for CI. Percentage in B minus percentage in C needed to be greater than non-inferiority margin of -20%

2. Secondary Outcome: Change in the Total Volume of the Three Largest Myomas From Baseline to Week 13
Description: Assessment of PGL4001 capacity to decrease volume of the three largest myomas was performed at each center by means of ultrasonography at baseline and at week 13.
  The total volume of the three largest myomas assessed at screening and at end-of-treatment visit (Week 13) was analysed on a logarithm transformed scale (to base 10).
Time Frame: 3 months
Population: Per protocol
Measure: Mean (Standard Error); unit: Log 10 (Log cm3) Total volume
Arm/Group | A (PGL4001 5mg) | B (PGL4001 10mg) | C (GnRH-agonist)
Number analyzed (Participants) | 89 | 91 | 91
Log 10 (Log cm3) Total volume | -0.179 (0.037) [-58 to -11] | -0.220 (0.036) [-69 to -14] | -0.268 (0.037) [-69 to -36]
Statistical Analysis 1: Comparison: A (PGL4001 5mg) vs C (GnRH-agonist); Test type: Non-Inferiority or Equivalence — Non-inferiority; ANCOVA — No p-values generated; Analysis of covariance after log transformation of the data; Mean Difference (Final Values) = 0.089, 95% CI 2-sided [-0.003 to 0.181] — As comparison of 2 doses of PGL4001 vs GnRH-agonist, Bonneferroni correction used to adjust confidence intervals
Statistical Analysis 2: Comparison: B (PGL4001 10mg) vs C (GnRH-agonist); Test type: Non-Inferiority or Equivalence — Non-inferiority; ANCOVA — No p-values generated; Analysis of covariance after log transformation of the data; Mean Difference (Final Values) = 0.049, 95% CI 2-sided [-0.043 to 0.14] — As comparison of 2 doses of PGL4001 vs GnRH-agonist, Bonneferroni correction used to adjust confidence intervals

3. Primary Outcome: Co-primary Safety Endpoint: Serum Estradiol Levels at End of Treatment Visit (Week 13 Visit) for PGL4001 Compared With GnRHagonist
Description: Measured by log 10 (log pg/ml) transformed values for estradiol (E2) in blood samples
Time Frame: Week 13 visit
Population: Safety population
Measure: Mean (Standard Error); unit: log 10 (log pg/ml) E2
Arm/Group | A (PGL4001 5mg) | B (PGL4001 10mg) | C (GnRH-agonist)
Number analyzed (Participants) | 97 | 103 | 101
log 10 (log pg/ml) E2 | 1.897 (0.041) [45.0 to 110.0] | 1.843 (0.041) [35.0 to 121.0] | 1.381 (0.041) [10.0 to 36.0]
Statistical Analysis 1: Comparison: A (PGL4001 5mg) vs C (GnRH-agonist); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Since comparisons of 2 doses of ulipristal acetate vs GnRH-agonist, Bonferroni correction was used, p values were doubled (p-value threshold was 0.05) and CI adjusted; Analysed via Cochran-Mantel-Haenszel test, controlling for strata; Mean Difference (Net) = -28.3, 95% CI 2-sided [-40.6 to -14.6]
Statistical Analysis 2: Comparison: B (PGL4001 10mg) vs C (GnRH-agonist); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 3, analysis 1]; Analysed via Cochran-Mantel-Haenszel test, controlling for strata; Mean Difference (Net) = -29.9, 95% CI 2-sided [-42.0 to -16.6]

4. Primary Outcome: Co-primary Safety Endpoint: % of Subjects Reporting Moderate or Severe Hot Flushes as Adverse Events Throughout the Treatment Period for PGL4001 Compared With GnRH-agonist
Description: Difference in percentage of subjects reporting moderate or severe hot flushes:
  Frequency and severity of this adverse event(as spontaneously reported by patients or elicited by nonleading questions) were recorded on standard forms at every visit up to week 17.
Time Frame: Up to week 17
Population: Safety population
Measure: Number; unit: percentage of patients
Arm/Group | A (PGL4001 5mg) | B (PGL4001 10mg) | C (GnRH-agonist)
Number analyzed (Participants) | 97 | 103 | 101
percentage of patients | 11.3 [-40.6 to -14.6] | 9.7 [-42.0 to -16.6] | 39.6
Statistical Analysis 1: Comparison: A (PGL4001 5mg) vs C (GnRH-agonist); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Since planned analyses involved comparisons of 2 doses of PGL4001 vs GnRH-agonist, a Bonferroni correction was used and p values were doubled (p-value threshold was 0.05) and confidence intervals were similarly adjusted; Analysed via a Cochran-Mantel-Haenszel test, controlling for strata; Mean Difference (Net) = -28.3, 95% CI 2-sided [-40.6 to -14.6]
Statistical Analysis 2: Comparison: B (PGL4001 10mg) vs C (GnRH-agonist); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Analysed via a Cochran-Mantel-Haenszel test, controlling for strata; Median Difference (Net) = -29.9, 95% CI 2-sided [-42.0 to -16.6]

ADVERSE EVENTS:
Arm/Group | A (PGL4001 5mg) | B (PGL4001 10mg) | C (GnRH-agonist)
Serious Adverse Events (participants affected / at risk) | 5/97 | 4/103 | 4/101
Other Adverse Events (participants affected / at risk) | 75/97 | 79/103 | 85/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A (PGL4001 5mg) (N=97) | B (PGL4001 10mg) (N=103) | C (GnRH-agonist) (N=101)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Operative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Uterine hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Hemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Choriomeningitis lymphocytic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A (PGL4001 5mg) (N=97) | B (PGL4001 10mg) (N=103) | C (GnRH-agonist) (N=101)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 39 (50) | 44 (61) | 70 (103)
Hot flush (Reproductive system and breast disorders) | 25 (26) | 25 (26) | 66 (79)
Dysmenorrhea (Reproductive system and breast disorders) | 4 (6) | 5 (5) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 3 (4) | 5 (5) | 3 (3)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 5 (5) | 2 (3)
Breast pain (Reproductive system and breast disorders) | 4 (4) | 1 (1) | 2 (2)
Nervous system disorders (Nervous system disorders) | 30 (47) | 27 (33) | 34 (62)
Headache (Nervous system disorders) | 25 (38) | 19 (24) | 29 (49)
Migraine (Nervous system disorders) | 2 (3) | 3 (3) | 3 (6)
Gastrointestinal disorders (Gastrointestinal disorders) | 17 (19) | 21 (33) | 22 (35)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 9 (10) | 9 (9)
Nausea (Gastrointestinal disorders) | 6 (6) | 7 (7) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 3 (3) | 5 (7)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (5)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4)
Infections and infestations (Infections and infestations) | 14 (20) | 16 (19) | 16 (23)
Nasopharyngitis (Infections and infestations) | 6 (6) | 4 (4) | 2 (2)
Influenza (Infections and infestations) | 2 (2) | 2 (2) | 5 (5)
Pharyngitis (Infections and infestations) | 5 (5) | 0 (0) | 2 (2)
Vaginal infection (Infections and infestations) | 0 (0) | 2 (2) | 3 (3)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 12 (13) | 17 (18) | 12 (15)
Procedural pain (Injury, poisoning and procedural complications) | 9 (10) | 15 (15) | 9 (12)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 8 (10) | 13 (15) | 10 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (3)
General disorders and administration site conditions (General disorders) | 7 (7) | 17 (21) | 9 (11)
Fatigue (General disorders) | 4 (4) | 7 (8) | 3 (3)
Asthenia (General disorders) | 0 (0) | 4 (4) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 5 (5) | 11 (12) | 13 (14)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (6) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Psychiatric disorders (Psychiatric disorders) | 4 (5) | 4 (6) | 13 (15)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2) | 5 (5)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 6 (6) | 3 (3) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 3 (3) | 5 (5)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 6 (6) | 3 (3) | 4 (4)
Hypercholesterolemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 1 (1)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 4 (4) | 5 (5) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 5 (5) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No